CLINICAL TRIAL: NCT01572246
Title: Effects of Surgical Monopolar Electrocautery and Optimal Electrosurgery Unit Return Pad Placement on Implantable Cardioverter Defibrillators Protocol
Brief Title: Effects of Monopolar Electrocautery Use During Surgery on Implanted Cardiac Defibrillators
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Peter Schulman, Assistant Professor, Oregon Health and Science University
Other Study IDs: ISROTH20028
Record Dates: First submitted 2012-03-27; First posted 2012-04-06 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2016-08

CONDITIONS: Heart Failure; Tachycardia, Ventricular
Keywords: electrosurgery; Cardiac surgical procedures; Surgical procedures, operative; Defibrillators
MeSH Terms: conditions — Heart Failure; Tachycardia, Ventricular; Hyperthermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Non-cardiac above-the-waist surgery: Subjects with an implanted ICD who present for a non-cardiac above-the-waist surgical procedure involving monopolar electrocautery
  Interventions: Other: Optimal placement of return pad
- Cardiac surgery: Subjects with an implanted ICD who present for a cardiac surgical procedure involving monopolar electrocautery
- Below-the-waist surgery: Subjects with an implanted ICD who present for a below-the-waist surgical procedure involving monopolar electrocautery

INTERVENTIONS:
Other: Optimal placement of return pad — The ESU return pad will be placed in an optimal position in order to direct ME current away from the ICD pulse generators.
  Groups: Non-cardiac above-the-waist surgery

SUMMARY:
This observational protocol will evaluate the effects of monopolar electrocautery (ME) on implantable cardioverter defibrillators (ICDs) in patients undergoing surgery. ME can cause electromagnetic interference (EMI) leading to ICD damage or inadvertent ICD discharge (shocks). Recommended practice calls for the preoperative reprogramming of ICDs when ME will be used to prevent patients from receiving inadvertent shocks. This requires the presence of someone trained in ICD programming, but a trained person is not always readily available.

In this study the investigators will reprogram ICDs prior to surgery according to current practice, but will also record what would have happened had the ICD reprogramming not occurred ("detection on" but "therapy off"). In addition, the investigators will evaluate the effect of the location of the electrosurgery unit (ESU) return pad on the incidence of EMI. The investigators hypothesize that directing the current return path away from the ICD will result in lower EMI rates than previously described.

ELIGIBILITY:
Inclusion Criteria:

* Adult individuals of both genders, 18 years of age and older
* For patients undergoing surgery about the waist, previous implantation of a functioning Boston Scientific or Medtronic ICD
* For patients undergoing surgery below the waist, previous implantation of a functioning Boston Scientific, Medtronic, St. Jude Medical, or Biotronik ICD
* Signed informed consent

Exclusion Criteria:

* Surgery involving the ICD pocket (generator change out procedure)
* Surgery or procedures exclusively involving bipolar electrocautery (such as ophthalmic surgery)
* Patients undergoing surgery above the waist with ICDs not manufactured by Medtronic or Boston Scientific (other ICDs do not allow reprogramming to allow EMI detection without the potential for inadvertent ICD discharge)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with ICDs (including cardiac resynchronization therapy system-defibrillators) scheduled for surgery involving ME.
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2012-05; Primary Completion 2016-09-14 (Actual); Study Completion 2016-09-14 (Actual)

PRIMARY OUTCOMES:
Incidence of electromagnetic interference (EMI) | During surgery on day of enrollment
  Evaluation of occurence of EMI when monopolar electrocautery is used in surgical procedures when the patient has an existing ICD.

SECONDARY OUTCOMES:
Incidence of unexpected preoperative ICD-related problems | Up to 6 months prior to date of surgery
  Determine the incidence and nature of unexpected preoperative ICD-related problems, such as inadequate pacing or sensing thresholds, battery at or near elective replacement interval, and lead fracture, as detected by preoperative ICD interrogation.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schulman, MD, Principal Investigator — Oregon Health and Science University; Charles Henrikson, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Background] American Society of Anesthesiologists. Practice advisory for the perioperative management of patients with cardiac implantable electronic devices: pacemakers and implantable cardioverter-defibrillators: an updated report by the american society of anesthesiologists task force on perioperative management of patients with cardiac implantable electronic devices. Anesthesiology. 2011 Feb;114(2):247-61. doi: 10.1097/ALN.0b013e3181fbe7f6. No abstract available. PMID 21245737
- [Background] Crossley GH, Poole JE, Rozner MA, Asirvatham SJ, Cheng A, Chung MK, Ferguson TB Jr, Gallagher JD, Gold MR, Hoyt RH, Irefin S, Kusumoto FM, Moorman LP, Thompson A. The Heart Rhythm Society (HRS)/American Society of Anesthesiologists (ASA) Expert Consensus Statement on the perioperative management of patients with implantable defibrillators, pacemakers and arrhythmia monitors: facilities and patient management this document was developed as a joint project with the American Society of Anesthesiologists (ASA), and in collaboration with the American Heart Association (AHA), and the Society of Thoracic Surgeons (STS). Heart Rhythm. 2011 Jul;8(7):1114-54. doi: 10.1016/j.hrthm.2010.12.023. No abstract available. PMID 21722856
- [Background] Stone KR, McPherson CA. Assessment and management of patients with pacemakers and implantable cardioverter defibrillators. Crit Care Med. 2004 Apr;32(4 Suppl):S155-65. doi: 10.1097/01.ccm.0000115622.73988.6e. PMID 15064674
- [Background] Rozner MA. The patient with a cardiac pacemaker or implanted defibrillator and management during anaesthesia. Curr Opin Anaesthesiol. 2007 Jun;20(3):261-8. doi: 10.1097/ACO.0b013e32814f1c4a. PMID 17479032
- [Background] Korantzopoulos P, Letsas KP, Grekas G, Goudevenos JA. Pacemaker dependency after implantation of electrophysiological devices. Europace. 2009 Sep;11(9):1151-5. doi: 10.1093/europace/eup195. Epub 2009 Jul 16. PMID 19617204
- [Background] Cheng A, Nazarian S, Spragg DD, Bilchick K, Tandri H, Mark L, Halperin H, Calkins H, Berger RD, Henrikson CA. Effects of surgical and endoscopic electrocautery on modern-day permanent pacemaker and implantable cardioverter-defibrillator systems. Pacing Clin Electrophysiol. 2008 Mar;31(3):344-50. doi: 10.1111/j.1540-8159.2008.00996.x. PMID 18307631
- [Background] Fiek M, Dorwarth U, Durchlaub I, Janko S, Von Bary C, Steinbeck G, Hoffmann E. Application of radiofrequency energy in surgical and interventional procedures: are there interactions with ICDs? Pacing Clin Electrophysiol. 2004 Mar;27(3):293-8. doi: 10.1111/j.1540-8159.2004.00430.x. PMID 15009852
- [Background] Antiarrhythmics versus Implantable Defibrillators (AVID) Investigators. A comparison of antiarrhythmic-drug therapy with implantable defibrillators in patients resuscitated from near-fatal ventricular arrhythmias. N Engl J Med. 1997 Nov 27;337(22):1576-83. doi: 10.1056/NEJM199711273372202. PMID 9411221
- [Background] Moss AJ, Zareba W, Hall WJ, Klein H, Wilber DJ, Cannom DS, Daubert JP, Higgins SL, Brown MW, Andrews ML; Multicenter Automatic Defibrillator Implantation Trial II Investigators. Prophylactic implantation of a defibrillator in patients with myocardial infarction and reduced ejection fraction. N Engl J Med. 2002 Mar 21;346(12):877-83. doi: 10.1056/NEJMoa013474. Epub 2002 Mar 19. PMID 11907286